CLINICAL TRIAL: NCT00311844
Title: A Double-blind, Placebo-controlled, Crossover, Single-center Study to Evaluate the Anti-allergic and Anti-inflammatory Effects of Multiple Doses of Desloratadine on Conjunctival Allergen Challenge-induced Ocular Signs and Symptoms
Brief Title: A Study of the Effects of Desloratadine on Conjunctival Allergen Challenge-induced Ocular Signs and Symptoms (Study P04209)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P04209
Record Dates: First submitted 2006-04-04; First posted 2006-04-06 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Conjunctivitis, Allergic
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — desloratadine

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: desloratadine

SUMMARY:
This study was a double-blind, placebo-controlled, cross-over, single-center study of desloratadine 5 mg or placebo in subjects 18 years of age or older with a history of seasonal allergic rhinoconjunctivitis. This study was performed to examine the effects of desloratadine compared with placebo, on the signs and symptoms of allergic conjunctivitis induced by direct conjunctival challenges with a previously identified sensitizing antigen, in the eyes of a subject known to be sensitive to the antigen.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study and comply with the procedures, including adherence to dosing and visit schedules by signing informed consent
* 18 years of age or older, of either sex, and race, with normal health and asymptomatic
* At least a 2-year history (self-reported acceptable) of recurrent seasonal allergic conjunctivitis associated with seasonal allergic rhinitis
* Skin test positive (skin prick test with a wheal diameter at least 3 mm larger than the diluent control or intradermal testing with the wheal diameter at least 7 mm larger than diluent control) at Screening, or within 12 months prior to the Screening Visit, to an appropriate seasonal allergen, including one or more of the following: Kentucky bluegrass (Poa pratensis)grass: meadow fescue, rye, Bermuda grass trees: oak, maple, birch cat hair or dander (Felis domesticus) ragweed
* Female subjects of childbearing potential must be using an acceptable method of birth control (ie, hormonal contraceptive, medically prescribed IUD, condom in combination with spermicide) or be surgically sterilized
* Female subjects of childbearing potential must have a negative urine pregnancy test at the Screening Visit
* A calculated best-corrected visual acuity of 0.6 logMar or better in each eye as measured by an ETDRS chart
* Free of any clinically significant disease (other than SAR) that would interfere with study evaluations.
* Must agree to record symptom severity scores, medication times, concomitant medications, and adverse events accurately and consistently in a daily diary.
* At the Screening Visit, prior to the qualifying conjunctival allergen challenge, the subject must have an ocular symptom severity redness score of mild (<=1) prior to exposure to allergen. Following allergen challenge, the subject must achieve ocular itching and redness scores of at least moderate (>=2) in both eyes within 10 minutes of the last allergen challenge. For redness, the score must be >=2 in 2 of the 3 vessel beds. (details in section 8.2.6 and 8.3.2 of the protocol)
* At the confirmation visit, the subject must have ocular itching scores in both eyes of >=2 in 2 of the 3 timepoints (3, 5, and 7 minutes post-challenge). The subject must also have the following redness score bilaterally at 15 minutes post-challenge: >=2 in at least 2 vessel beds and >=6 composite oculare redness score

Exclusion Criteria:

* A female who is pregnant, intends to become pregnant during the study or is nursing
* Subject has not observed the designated washout periods for prohibited medication as per protocol Section 7.2. Antihistamines, inhaled nasal cromones, and inhaled nasal corticosteroids are prohibited for the months

prior to Screening Visit

* Current evidence of clinically significant hematopoietic, cardiovascular, hepatic, immunologic, renal, neurologic, psychiatric, autoimmune disease or other disease including those that would interfere with the absorption, distribution, metabolism, or excretion of the study drug, or with the subject's ability to complete diary cards
* Clinically significant deviation from normal in the physical and ocular exam, which may interfere with study evaluation or affect subject safety
* Participation in another clinical study
* Use of any investigational product within 30 days of enrollment
* Subject is part of the study staff or family member of the staff directly involved with this study
* History of asthma being treated with inhaled or oral corticosteroids, beta-2-agonists, cromones, theophylline, or leukotriene inhibitors and cannot complete washout and study period without these medications
* A respiratory or ocular infection during the 4 weeks prior to pre-dose evaluations
* History of intranasal drug abuse
* Known potential for hypersensitivity, allergy or idiosyncratic reaction to study drug or excipients, or Claritin
* Upper respiratory tract or sinus infection that required antibiotics within 28 days of Screening, or had a viral upper respiratory infection within 7 days of Screening, or has persistent symptoms at Screening Visit
* Dependence on nasal, oral, or ocular decongestants, nasal topical antihistamines or nasal steroids
* Subjects on immunotherapy must remain on stable dose during the study. Subjects are not to have received desensitization treatment within 24 hours prior to a visit
* History of non-compliance with medication or treatment protocols
* History of difficulty swallowing pills or has known upper gastrointestinal narrowing or abnormal esophageal peristalsis
* Subject is a night-shift worker or does not have standard asleep at night/awake during the day cycle
* Unwilling to discontinue use of contact lenses during the course of the study
* Subject's ability to provide informed consent is compromised

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2005-03-01 (Actual); Primary Completion 2005-05-28 (Actual); Study Completion 2005-05-28 (Actual)

REFERENCES:
- [Result] Torkildsen GL, Gomes P, Welch D, Gopalan G, Srinivasan S. Evaluation of desloratadine on conjunctival allergen challenge-induced ocular symptoms. Clin Exp Allergy. 2009 Jul;39(7):1052-9. doi: 10.1111/j.1365-2222.2009.03224.x. Epub 2009 Mar 10. PMID 19302250